CLINICAL TRIAL: NCT05050617
Title: Point-of-Care Ultrasound in Predicting Adverse Outcomes in Emergency Department Patients With Acute Pulmonary Embolism
Status: Recruiting | Type: Observational
Sponsor: WellSpan Health (Other)
Collaborators: Stony Brook University (Other); University of California, Irvine (Other)
Responsible Party: Principal Investigator, Brent Becker, Research Director, Department of Emergency Medicine, WellSpan Health
Other Study IDs: 1793729-1
Record Dates: First submitted 2021-08-31; First posted 2021-09-20 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute Pulmonary Embolism: Subjects in this single cohort will undergo point-of-care echocardiography at the time of presentation and subsequent follow up to assess for short term adverse events or complications.
  Interventions: Diagnostic Test: Point-of-care echocardiography

INTERVENTIONS:
Diagnostic Test: Point-of-care echocardiography — Subjects will undergo point-of-care echocardiography at the time of presentation/enrollment to assess for evidence of right sided heart dilation/strain.

SUMMARY:
This study is an observational, prospective study examining the role point-of-care echocardiography of predicting short term adverse outcomes in emergency department patients with acute pulmonary embolism.

The primary objective is to assess the diagnostic performance of ultrasound-guided measures of right ventricular dilation (RVD) and strain in predicting clinical outcomes in acute PE.

The secondary objective is to investigate the utility of combining ultrasound-guided measures of RVD and the pulmonary embolism severity index (PESI) score in predicting adverse outcomes in acute PE.

DETAILED DESCRIPTION:
STUDY: Point-of-Care Ultrasound in Predicting Adverse Outcomes in Emergency Department Patients With Acute Pulmonary Embolism

BACKGROUND

The clinical outcomes associated with pulmonary embolism (PE) vary widely. In the United States, most patients are admitted for inpatient therapy; however, there is evidence to suggest that outpatient therapy may be safe in patients with non-massive PEs. Appropriate outpatient treatment of patients with pulmonary emboli not only has the potential to increase patient satisfaction, but also has the potential to significantly reduce cost of care without compromising patient safety.

The pulmonary embolism severity index (PESI) is an externally validated prediction tool for mortality associated with PE. The PESI consists of 11 clinical parameters that are routinely available and stratifies patients into 5 risk categories, class I having the lowest risk of short-term mortality and class V having the highest. The PESI does not rely on imaging modalities to determine risk of adverse outcome within 30 days of initial PE diagnosis.

Predicting short-term adverse outcomes in PE is essential for proper disposition, namely hospitalization of at-risk patients and discharge of those with low likelihood of decompensation. Hariharan et al. evaluated the ability of PESI to predict short-term deterioration (<5 days) in patients with acute PE. The PESI demonstrated a sensitivity of 86% (95% CI 73-93%) for predicting short-term adverse events. Approximately 14% of patients deemed low-risk by PESI required short-term interventions. The authors concluded that risk stratification with PESI warrants further optimization.

Further research in South Korea has suggested combining CT findings of right ventricular dysfunction (RVD) with the PESI score improved predictive accuracy. Right heart strain may be an independent prognostic factor of adverse outcomes in patients with acute PE, and may enhance prognosis versus PESI score alone.

Point-of-care (POC) echocardiography has been shown to be a useful diagnostic tool to detect RVD. Several parameters can provide morphological, functional, and hemodynamic information that are obtainable using a bedside study. These include tricuspid annular plane systolic excursion (TAPSE) and 60/60 sign.

POC ultrasound (US) can be performed at the bedside by trained emergency physicians to assess for these markers of RVD. The investigators hypothesize this will yield significant benefit in risk stratifying individuals with acute PE and potentially influence disposition. This study aims to assess the role of US-guided measures of RVD in predicting clinical outcomes in patients with acute PE, both in isolation and in conjunction with PESI scores.

OBJECTIVES

1. To assess the diagnostic performance of ultrasound-guided measures of RVD, specifically TAPSE and the 60-60 sign, in predicting short term clinical outcomes in acute PE
2. To investigate the diagnostic performance of combining ultrasound-guided measures of RVD (TAPSE and 60-60 sign) and the PESI score in predicting short term adverse outcomes in acute PE

RESEARCH METHODS

Study Design

This is an observational, prospective study of patients presenting to the ED and diagnosed with acute PE by CT imaging. Screening for potential subjects will be conducted by ED staff working clinically, as well as ultrasound/procedure emergency medicine residents and US fellows/faculty on "scanning shifts". Informed consent will be obtained by a member of the study team prior to data collection or study procedures. A POC ultrasound will be performed by an ED attending, fellow or resident under the supervision of an emergency physician accredited in bedside echocardiography, which is considered standard of care. Data regarding the initial presentation, components of the PESI score and POC ultrasound will be documented at the bedside. Ultrasound images will be recorded via the usual ultrasound archival software and undergo the standard QA process. ED residents/fellows/attendings participating in this study will be trained on study protocols by accredited staff prior to participation in consent, ultrasonography and data collection.

Patients enrolled in the study will receive telephone follow-up calls from the research team at 7 (+/- 3) and 30 (+/- 5) days from the date of PE diagnosis. Questions will focus on subsequent adverse outcomes, including development of recurrent PE/DVT, new cardiac dysrhythmia, advanced cardiac life support, advanced respiratory support, need for pressor support, need for thrombolysis, development of major bleeding, return to the ED, or death.

Additional follow up data will be collected via review of the electronic medical record and documented on a standardized data collection form after 30 days from initial diagnosis.

Study Population and Recruitment Methods

Study population will include ED patients over the age of 18 who are identified as have an acute pulmonary embolism on CT imaging. Patients will be seen initially by the treating physician and receive the usual standard of care. If an acute PE is identified, the treating physician will contact a member of the study team to assess eligibility, discuss the study with the patient and obtain consent. The POC ultrasound may be performed by a physician member of the study team or another credentialed emergency physician.

Role of Subjects

The study subjects will receive standard treatment at the discretion of the treating physician and resident team. The patient's decision to participate in this study will not directly affect their care in the ED. The treating physician and resident team will not necessarily be blinded to the findings of the POC US as this may yield important clinical information.

Research Procedures

Screening for inclusion in this study will occur in the Emergency Department as outlined above. Informed consent will be given to eligible patients for review. Written informed consent will be obtained prior to ultrasound imaging. Ultrasound images will be saved and stored securely on the hospital server. Ultrasonographic findings and initial clinical data will be recorded on a Bedside Standardized Data Collection Form during the exam. Follow up clinical information from chart review and telephone calls will be recorded on a Follow Up Standardized Data Collection Form.

Each patient will be assigned a study ID number at the time of enrollment and a linking document will be maintained. Once data collection is complete, forms will be de-identified by the removal of the patient's name/MRN/FIN/identifying information.

Ultrasound Technique

All POC echocardiograms will be obtained utilizing 2.5-3.5 MHz transducers by a credentialed physician sonographer during initial evaluation in the ED. Patients will be examined in the supine or left lateral decubitus position.

TAPSE serves as a quantitative measure of right heart dysfunction. TAPSE will be calculated by obtaining a standard apical four chamber view with M-mode placed over the lateral tricuspid annulus to measure the maximal excursion of the RV between the end of diastole to the end of systole. Patients will be divided into high risk, moderate risk, and low risk groups based on TAPSE measurements of <16 mm, 16-20 mm, and >20 mm respectively.

60/60 sign is defined as both a pulmonary artery systolic pressure (PASP) of <60 mmHg and pulmonary acceleration time (PAT) of <60 msecs. In patients without chronic right heart remodeling, PASP can be estimated using right ventricular systolic pressures (RVSP). RVSP calculation relies on both estimating the tricuspid gradient (TG) and the right atrial pressure (RAP). Right atrial pressure in non-ventilated patients can be approximated using central venous pressure. By placing the ultrasound probe in sagittal axis subxiphoid view, the IVC size can be measured at 2 cm distal to the right atrium. A plethoric IVC with a large diameter of >2.1 cm with <50% collapse with respiration estimates a RAP of 15 mmHg, which is considered elevated. A diameter of >2.1 cm with >50% collapse or a diameter of <2.1 cm with <50% collapse estimates a RAP of 8 mmHg, which is considered normal. A narrow IVC with a diameter of <2.1 cm and >50% collapse with respiratory variation estimates a RAP of 3 mmHg. (10) TG is measured using tricuspid regurgitation jet. While using standard apical 4 chamber view, color flow will be applied across the tricuspid valve to identify regurgitation jet. Continuous wave doppler will be applied in the middle of the jet. Peak blood flow (TRmax) will be measured at the apex of the waveform.

TG will then be calculated using the equation:

TG = 4 x (TRmax) 2

RVSP will be calculated using the equation:

RVSP = TG + RAP

An RVSP of <60 mmHg suggests acute RV dysfunction whereas an RVSP of >60 mmHg suggests chronic RV dysfunction.

PAT refers to the amount of time it takes to reach peak pulmonic velocity. PAT will be calculated using the basal short axis view with power Doppler aligned with blood flow through the pulmonic valve with sweep speed increased to measure the time between the initial blood flow to peak blood flow. A PAT of <60 msecs indicates that the pulmonic velocity and pressure peak very quickly, suggesting an acute cause of RV dysfunction. (4, 10)

Data Analysis/Sample Size Calculations

Descriptive statistics will be reported as means/medians with standard deviations/interquartile ranges for continuous variables and proportions with percentages for categorical variables. The diagnostic performance of PESI score, POC echocardiography and the combination of PESI+POC echocardiography for predicting the primary and secondary outcomes will be calculated, including sensitivity, specificity, likelihood ratios, and negative/positive predictive values (NPV/PPV) with associated 95% confidence intervals. Interrater reliability for follow up data collection from the medical record will be assessed via Cohen's Kappa. p<0.05 will be considered statistically significant.

The investigators anticipate approximately 30% of the enrolled acute PE population will experience at least one component of the primary composite outcome. Setting a goal sensitivity of 95% (+/- 5%) for the combined PESI+POC echocardiography prediction tool, assuming alpha=0.05, beta=0.2 and allowing for an approximated 10% attrition rate, the investigators estimate that 250 patients will be required to achieve adequate statistical power.

Risks and Risk Management

There are minimal risks to patients participating in this study since ultrasound is non-invasive and known to be safe. There is a slight risk of the participants' privacy or confidentiality being breached. Standard precautions will be taken to ensure privacy and confidentiality is maintained during the study.

Benefits

Subjects may receive clinical benefit from the additional information provided by POC echocardiography; however, the disposition and treatment of patients enrolled in this study will remain at the discretion of the primary attending and resident team. The results of the ultrasound study will be made available to the clinical team.

Alternative Procedures

Patients who decline to participate in the study will not have the quality of their treatment affected in any way.

Research materials, records, confidentiality

Research records will be stored in locked offices, filing cabinets, and computers using passwords.

Subject informed consent

We will seek documented informed consent and HIPAA Authorization. Patients who decline participation will continue their usual treatment course in the ED.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years of age
* ED diagnosis of acute pulmonary embolism with identification on CT imaging

Exclusion Criteria:

* Age <18 years of age
* Inability to provide informed consent
* Incarceration
* Current PE previously diagnosed prior to index ED visit

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population consists of ED patients over the age of 18 who have an acute pulmonary embolism identified on CT imaging.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2021-09-09 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Adverse Events at 5 days | Within 5 days of presentation/enrollment
  Composite of recurrent/worsening VTE (including PE or DVT), new cardiac dysrhythmia, major bleeding, return to the ED, death or need for critical interventions (including advanced cardiac life support, advanced respiratory support, vasopressor support, thrombolysis or new oxygen requirement occurring after initial presentation) occurring within 5 days of acute PE diagnosis

SECONDARY OUTCOMES:
Adverse Events during Index Hospitalization | Between time of presentation/enrollment and discharge from index hospitalization
  Composite of mortality, major bleeding or recurrent/worsening PE during index hospitalization
Adverse Events within 14 days | Within 14 days of presentation/enrollment
  Composite of mortality, major bleeding or recurrent/worsening PE within 14 days of presentation/enrollment
Adverse Events within 30 days | Within 30 days of presentation/enrollment
  Composite of mortality, major bleeding or recurrent/worsening PE within 30 days of presentation/enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Brent A Becker, MD, Principal Investigator — WellSpan Health
Locations (1):
- Wellspan York Hospital, York, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Alerhand S, Hickey SM. Tricuspid Annular Plane Systolic Excursion (TAPSE) for Risk Stratification and Prognostication of Patients with Pulmonary Embolism. J Emerg Med. 2020 Mar;58(3):449-456. doi: 10.1016/j.jemermed.2019.09.017. Epub 2019 Nov 15. PMID 31735658
- [Background] Aujesky D, Perrier A, Roy PM, Stone RA, Cornuz J, Meyer G, Obrosky DS, Fine MJ. Validation of a clinical prognostic model to identify low-risk patients with pulmonary embolism. J Intern Med. 2007 Jun;261(6):597-604. doi: 10.1111/j.1365-2796.2007.01785.x. PMID 17547715
- [Background] Carley S, Dosman S, Jones SR, Harrison M. Simple nomograms to calculate sample size in diagnostic studies. Emerg Med J. 2005 Mar;22(3):180-1. doi: 10.1136/emj.2003.011148. PMID 15735264
- [Background] Chan CM, Woods C, Shorr AF. The validation and reproducibility of the pulmonary embolism severity index. J Thromb Haemost. 2010 Jul;8(7):1509-14. doi: 10.1111/j.1538-7836.2010.03888.x. Epub 2010 Apr 16. PMID 20403093
- [Background] Ciurzynski M, Kurnicka K, Lichodziejewska B, Kozlowska M, Plywaczewska M, Sobieraj P, Dzikowska-Diduch O, Goliszek S, Bienias P, Kostrubiec M, Pruszczyk P. Tricuspid Regurgitation Peak Gradient (TRPG)/Tricuspid Annulus Plane Systolic Excursion (TAPSE) - A Novel Parameter for Stepwise Echocardiographic Risk Stratification in Normotensive Patients With Acute Pulmonary Embolism. Circ J. 2018 Mar 23;82(4):1179-1185. doi: 10.1253/circj.CJ-17-0940. Epub 2018 Jan 26. PMID 29375106
- [Background] Daley J, Grotberg J, Pare J, Medoro A, Liu R, Hall MK, Taylor A, Moore CL. Emergency physician performed tricuspid annular plane systolic excursion in the evaluation of suspected pulmonary embolism. Am J Emerg Med. 2017 Jan;35(1):106-111. doi: 10.1016/j.ajem.2016.10.018. Epub 2016 Oct 11. PMID 27793505
- [Background] Donze J, Le Gal G, Fine MJ, Roy PM, Sanchez O, Verschuren F, Cornuz J, Meyer G, Perrier A, Righini M, Aujesky D. Prospective validation of the Pulmonary Embolism Severity Index. A clinical prognostic model for pulmonary embolism. Thromb Haemost. 2008 Nov;100(5):943-8. doi: 10.1160/th08-05-0285. PMID 18989542
- [Background] Hariharan P, Takayesu JK, Kabrhel C. Association between the Pulmonary Embolism Severity Index (PESI) and short-term clinical deterioration. Thromb Haemost. 2011 Apr;105(4):706-11. doi: 10.1160/TH10-09-0577. Epub 2011 Jan 12. PMID 21225095
- [Background] Kurzyna M, Torbicki A, Pruszczyk P, Burakowska B, Fijalkowska A, Kober J, Oniszh K, Kuca P, Tomkowski W, Burakowski J, Wawrzynska L. Disturbed right ventricular ejection pattern as a new Doppler echocardiographic sign of acute pulmonary embolism. Am J Cardiol. 2002 Sep 1;90(5):507-11. doi: 10.1016/s0002-9149(02)02523-7. PMID 12208411
- [Background] Rydman R, Soderberg M, Larsen F, Alam M, Caidahl K. d-Dimer and simplified pulmonary embolism severity index in relation to right ventricular function. Am J Emerg Med. 2013 Mar;31(3):482-6. doi: 10.1016/j.ajem.2012.09.016. Epub 2012 Nov 12. PMID 23154103
- [Background] Shafiq Q, Moukarbel GV, Gupta R, Hernandez DA, Khouri SJ. Practical echocardiographic approach for risk stratification of patients with acute pulmonary embolism. J Echocardiogr. 2016 Dec;14(4):146-155. doi: 10.1007/s12574-016-0306-4. Epub 2016 Aug 10. PMID 27510333